CLINICAL TRIAL: NCT00089557
Title: An Open-Label Extension Study of NGX-4010 for the Treatment of Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: NeurogesX (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: C114
Record Dates: First submitted 2004-08-06; First posted 2004-08-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Herpes Zoster; Neuralgia; Pain; HIV Infections; Peripheral Nervous System Diseases; Diabetic Neuropathies; Diabetes Mellitus; Polyneuropathies
Keywords: Dermal assessment; Pain assessment; Diary; Analgesics; Capsaicin; Herpes zoster; Neuralgia; Pain; HIV Infections; Peripheral Nervous System Diseases; Diabetic Neuropathies; Diabetes Mellitus; Polyneuropathies; Complementary Therapies
MeSH Terms: conditions — Herpes Zoster; Neuralgia; Pain; HIV Infections; Peripheral Nervous System Diseases; Diabetic Neuropathies; Diabetes Mellitus; Polyneuropathies

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
This study is an open-label, multicenter, extension study for subjects who completed NeurogesX Study C111 and received treatment with NGX-4010 (Capsaicin Patch) within 12 weeks (up to +7days) before entry into Study C114

ELIGIBILITY:
Key Eligibility Criteria:

* Must have completed NeurogesX Study C111 and received treatment with NGX-4010 (Capsaicin Patch) within 12 weeks (up to +7 days) before entry into Study C114.
* Demonstrated adherence to protocol requirements during Study C111, and willing and able to comply with protocol requirements for the duration of the study participation.
* Must not have had any serious adverse experience since enrollment in Study C111, whether or not considered to be study drug-related.
* Must have intact skin at the treatment area.
* Must be prepared to remain on the same pain medications at the same doses as before the study for the entire duration of the study (36 weeks).
* Must not use topical pain medications on painful areas.
* Must be at least 18 years old, not pregnant, and able to take care of self independently, with only occasional assistance if needed.
* No history or current problem with substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult